CLINICAL TRIAL: NCT06461559
Title: Pilot Study of Preoperative Intestinal Training Using Antegrade Ileostomy Infusion
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Shanglei Liu, Assistant Professor of Surgery, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 810144
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-06

CONDITIONS: Stoma Ileostomy; Ileostomy; Complications

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Ileostomy infusion (Active Comparator): perform infusion if ileostomy prior to takedown operation
  Interventions: Device: antegrade infusion of ileostomy content

INTERVENTIONS:
Device: antegrade infusion of ileostomy content — infusing the contents of ileostomy output back into intestine of the patient
  Arms: Ileostomy infusion

SUMMARY:
This research study is being conducted to study the effect of infusing your contents from your ostomy bag back into your intestine to re-train them prior to the ostomy takedown operation, which is a surgery to reverse your ostomy to put your intestine back together. Because your intestine past the ostomy hasn't seen any intestinal content for several weeks to months before the takedown operation, it is no longer used to handling the daily work of processing intestinal content and will take time to recover its normal function after surgery. We hope to speed up this process by training them before your planned surgery.

ELIGIBILITY:
Inclusion Criteria:

* Has a diverting loop ileostomy
* undergoing evaluation for stoma takedown

Exclusion Criteria:

* unable to perform consent
* unable to perform stoma infusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
timing to return of bowel function | 1-5 days
  time to return of bowel function after stoma surgery

SECONDARY OUTCOMES:
ease of stoma infusion | 2 weeks prior to surgery to time of surgery
  how easy was it for patients to infuse contents
complications | 2 weeks prior to surgery to 30 days post operatively
  if there are any complications from using the stoma infusion

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided